CLINICAL TRIAL: NCT03351608
Title: A Phase 4 Double-Blinded, Randomized, Active Comparator-Controlled Clinical Trial to Study the Efficacy, Safety, and Pharmacokinetics of Sugammadex (MK-8616) for Reversal of Neuromuscular Blockade in Pediatric Participants
Brief Title: Efficacy, Safety, and Pharmacokinetics of Sugammadex for Reversal of Neuromuscular Blockade (NMB) in Pediatric Participants (MK-8616-089)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8616-089; 2017-000692-92 (EudraCT Number); MK-8616-089 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate; Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sugammadex 2 mg/kg (Part A) (Experimental): Single intravenous (i.v.) bolus of sugammadex at 2 mg/kg.
  Interventions: Drug: Sugammadex 2 mg/kg
- Sugammadex 4 mg/kg (Part A) (Experimental): Single i.v. bolus of sugammadex at 4 mg/kg.
  Interventions: Drug: Sugammadex 4 mg/kg
- Sugammadex 2 mg/kg (Part B) (Experimental): Single i.v. bolus of sugammadex at 2 mg/kg.
  Interventions: Drug: Sugammadex 2 mg/kg
- Sugammadex 4 mg/kg (Part B) (Experimental): Single i.v. bolus of sugammadex at 4 mg/kg.
  Interventions: Drug: Sugammadex 4 mg/kg
- Neostigmine (Part B) (Active Comparator): Single i.v. bolus containing neostigmine (50 μg/kg; up to 5 mg maximum dose) in combination with either glycopyrrolate (10 μg/kg) or atropine sulfate (20 μg/kg).
  Interventions: Drug: Neostigmine + Glycopyrrolate; Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: Sugammadex 2 mg/kg — For moderate NMB reversal, a single i.v. bolus of sugammadex (2 mg/kg) will be given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
  Other Names: MK-8616; BRIDION®
  Arms: Sugammadex 2 mg/kg (Part A); Sugammadex 2 mg/kg (Part B)
Drug: Sugammadex 4 mg/kg — For deep NMB reversal, a single i.v. bolus of sugammadex (4 mg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of detection of a target of 1 to 2 post-tetanic counts and no response to TOF stimulations (TOF=0).
  Other Names: MK-8616; BRIDION®
  Arms: Sugammadex 4 mg/kg (Part A); Sugammadex 4 mg/kg (Part B)
Drug: Neostigmine + Glycopyrrolate — For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as glycopyrrolate (10 μg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
  Arms: Neostigmine (Part B)
Drug: Neostigmine + Atropine — For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as atropine (20 μg/kg) will be given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
  Arms: Neostigmine (Part B)

SUMMARY:
This trial will evaluate the efficacy, safety, and pharmacokinetics of sugammadex for the reversal of both moderate and deep neuromuscular blockade (NMB) induced by either rocuronium or vecuronium in pediatric participants. The primary efficacy hypothesis of this investigation is that sugammadex is superior to neostigmine in reversing moderate NMB in pediatric participants as measured by time to recovery to a train-of-four (TOF) ratio of ≥0.9.

DETAILED DESCRIPTION:
This trial will be conducted in two parts: Part A and Part B. In Part A, pharmacokinetic (PK) sampling will be conducted to identify the pediatric dose providing sugammadex exposure similar to adults. For Part B participants, the efficacy of sugammadex (i.e. time to recovery of the TOF ratio) will be assessed. Further, safety analyses will be conducted in both Parts A and B. Following completion of Part A, an interim analysis (IA) of the PK and safety data will be performed. Once the appropriate doses are confirmed and safety data is assessed for the 2 doses of sugammadex, then Part B will commence.

ELIGIBILITY:
Inclusion Criteria:

* Be categorized as American Society of Anesthesiologists (ASA) Physical Status Class 1, 2, or 3.
* Have a planned non-emergent surgical procedure or clinical situation (e.g., intubation) that requires moderate or deep NMB with either rocuronium or vecuronium.
* Have a planned surgical procedure or clinical situation that would allow objective neuromuscular monitoring techniques to be applied with access to the arm for neuromuscular transmission monitoring.
* Age between 2 to <17 years at Visit 2.
* If female, may participate if she is not pregnant, not breastfeeding, and at least one of the following: 1) Not a woman of childbearing potential (WOCBP); or 2) A WOCBP who agrees to follow the study contraceptive guidance during the treatment period and for at least 7 days after the last dose of study treatment.

Exclusion Criteria:

* Has any clinically significant condition or situation (eg, anatomical malformation that complicates intubation) other than the condition being studied that, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
* Has a neuromuscular disorder that may affect NMB and/or trial assessments.
* Is dialysis-dependent or has (or is suspected of having) severe renal insufficiency (defined as estimated glomerular filtration rate (eGFR) <30 ml/min).
* Has or is suspected of having a family or personal history of malignant hyperthermia.
* Has or is suspected of having an allergy to study treatments or its/their excipients, to opioids/opiates, muscle relaxants or their excipients, or other medication(s) used during general anesthesia.
* Has received or is planned to receive toremifene and/or fusidic acid via IV administration within 24 hours before or within 24 hours after administration of study treatment.
* Has been previously treated with sugammadex or has participated in a sugammadex clinical trial.
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days of signing the informed consent/assent for this current trial.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (11):
  - Childrens Hospital Los Angeles ( Site 0030), Los Angeles, California
  - Lucille Packard Children's Hospital ( Site 0006), Palo Alto, California
  - Rady Children's Hospital-San Diego ( Site 0035), San Diego, California
  - Children's National Medical Center ( Site 0008), Washington D.C., District of Columbia
  - C.S. Mott Children's Hospital/ University of Michigan Medical center ( Site 0014), Ann Arbor, Michigan
  - Saint Peter's University Hospital [New Brunswick, NJ] ( Site 0009), New Brunswick, New Jersey
  - Duke University Medical Center ( Site 0019), Durham, North Carolina
  - The Children's Hospital of Philadelphia ( Site 0015), Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC ( Site 0005), Pittsburgh, Pennsylvania
  - Memorial Hermann Medical Center University of Texas Medical School ( Site 0038), Houston, Texas
  - West Virginia University ( Site 0043), Morgantown, West Virginia
- Sozialmedizinisches Zentrum Ost - Donauspital ( Site 0150), Vienna, Austria
- Belgium (2):
  - Universitaire Ziekenhuis Antwerpen - UZA ( Site 0200), Edegem
  - UZ Leuven Campus Gasthuisberg ( Site 0201), Leuven
- Rigshospitalet ( Site 0250), Copenhagen, Denmark
- New Childrens Hospital ( Site 0750), Helsinki, Finland
- Germany (6):
  - Diakovere Annastift gGmbH ( Site 0354), Hanover
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 0355), Marburg
  - Klinikum Rechts der Isar Technische Universitaet Muenchen ( Site 0350), München
  - St. Franziskus-Hospital ( Site 0352), Münster
  - Klinikum am Steinenberg Reutlingen ( Site 0351), Reutlingen
  - Josephs-Hospitals Warendorf ( Site 0353), Warendorf
- Spain (4):
  - Hospital Santa Lucia ( Site 0501), Cartagena
  - Hospital Universitario Nino Jesus ( Site 0503), Madrid
  - Hospital Universitario La Paz ( Site 0502), Madrid
  - Clinica Universitaria de Navarra ( Site 0500), Pamplona
- Turkey (Türkiye) (4):
  - Ankara Universitesi Tip Fakultesi ( Site 0551), Ankara
  - Uludag Universitesi Tip Fakultesi ( Site 0553), Bursa
  - Koc Universitesi Hastanesi ( Site 0555), Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0552), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Voss T, Wang A, DeAngelis M, Speek M, Saldien V, Hammer GB, Wrishko R, Herring WJ. Sugammadex for reversal of neuromuscular blockade in pediatric patients: Results from a phase IV randomized study. Paediatr Anaesth. 2022 Mar;32(3):436-445. doi: 10.1111/pan.14370. Epub 2021 Dec 17. PMID 34878707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants 2 to <17 years of age who are categorized as American Society of Anesthesiologists (ASA) Physical Class 1, 2, or 3 and had a planned medical and/or surgical procedure requiring moderate or deep neuromuscular blockade (NMB) with rocuronium (ROC) or vecuronium (VEC) that would allow for neuromuscular monitoring were recruited.
Groups:
- Part A: Sugammadex 2 mg/kg: For moderate NMB reversal, a single intravenous (i.v.) bolus of sugammadex (2 mg/kg) was given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to train-of-four (TOF) stimulations.
- Part A: Sugammadex 4 mg; Part B: Sugammadex 4 mg/kg: For deep NMB reversal, a single i.v. bolus of sugammadex (4 mg/kg) was given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of detection of a target of 1 to 2 post-tetanic counts and no response to TOF stimulations (TOF=0).
- Part B: Sugammadex 2 mg/kg: For moderate NMB reversal, a single i.v. bolus of sugammadex (2 mg/kg) was given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
- Part B: Neostigmine + (Glycopyrrolate or Atropine): For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as either glycopyrrolate (10 μg/kg) or atropine (20 µg/kg) was given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
Period: Overall Study
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Started | 19 | 23 | 35 | 176 | 35
Treated | 18 | 22 | 33 | 169 | 34
Completed | 18 | 21 | 32 | 168 | 33
Not Completed | 1 | 2 | 3 | 8 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 2 | 1
Not completed — Randomized by mistake, no treatment given | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Sugammadex 2 mg/kg: For moderate NMB reversal, a single intravenous (i.v.) bolus of sugammadex (2 mg/kg) is given after the final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
- Part A: Sugammadex 4 mg; Part B: Sugammadex 4 mg/kg: For deep NMB reversal, a single i.v. bolus of sugammadex (4 mg/kg) is given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of detection of a target of 1 to 2 post-tetanic counts and no response to TOF stimulations (TOF=0).
- Part B: Sugammadex 2 mg/kg: For moderate NMB reversal, a single i.v. bolus of sugammadex (2 mg/kg) is given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
- Part B: Neostigmine + (Glycopyrrolate or Atropine): For moderate NMB reversal, a single i.v. bolus containing both neostigmine (50 μg/kg; up to 5 mg maximum dose) as well as either glycopyrrolate (10 μg/kg) or atropine (20 µg/kg) is given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
- Total: Total of all reporting groups
Arm/Group | Part A: Sugammadex 2 mg/kg | Part A: Sugammadex 4 mg | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine) | Total
Number analyzed (Participants) | 19 | 23 | 35 | 176 | 35 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.1 (4.7) | 7.2 (5.0) | 7.9 (4.4) | 7.9 (4.4) | 8.7 (4.4) | 7.9 (4.4)
Age, Customized [Number; unit: Participants]
  Children (2-11 years) | 15 | 17 | 25 | 132 | 25 | 214
  Adolescents (12-17 years) | 4 | 6 | 10 | 44 | 10 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 20 | 95 | 18 | 156
  Male | 8 | 11 | 15 | 81 | 17 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 3 | 5 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 0 | 6
  White | 16 | 17 | 30 | 161 | 33 | 257
  More than one race | 2 | 1 | 0 | 4 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Dosing to Infinity (AUC0-∞) of Sugammadex [Part A]
Description: The AUCo-∞ for sugammadex, defined as the area under the plasma concentration versus time plot, was determined in each Part A arm.
Time Frame: 2 minutes (min), 15 min, 30 min, 60 min, 4-6 hours (hrs), and 10 hrs post-dose
Population: All participants with ≥5 post-dosing samples available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Groups:
- Part A: Sugammadex 2 mg (2 to <6 Years): Participants in Part A receiving sugammadex 2 mg and who are 2 to <6 years of age are included.
- Part A: Sugammadex 2 mg (6 to <12 Years): Participants in Part A receiving sugammadex 2 mg and who are 6 to <12 years of age are included.
- Part A: Sugammadex 2 mg (12 to <17 Years): Participants in Part A receiving sugammadex 2 mg and who are 12 to <17 years of age are included.
- Part A: Sugammadex 4 mg (2 to <6 Years): Participants in Part A receiving sugammadex 4 mg and who are 2 to <6 years of age are included.
- Part A: Sugammadex 4 mg (6 to <12 Years): Participants in Part A receiving sugammadex 4 mg and who are 6 to <12 years of age are included.
- Part A: Sugammadex 4 mg (12 to <17 Years): Participants in Part A receiving sugammadex 4 mg and who are 12 to <17 years of age are included.
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years)
Number analyzed (Participants) | 9 | 5 | 4 | 8 | 6 | 6
hr*μg/mL | 14.1 (19.4) | 18.8 (27.4) | 27.6 (58.0) | 26.9 (18.5) | 38.2 (73.0) | 49.2 (20.1)

2. Primary Outcome: Plasma Clearance (CL) of Sugammadex [Part A]
Description: The CL of sugammadex, defined as the rate of elimination relative to plasma concentration, was determined in each Part A arm.
Time Frame: 2 minutes (min), 15 min, 30 min, 60 min, 4-6 hours (hrs), and 10 hrs post-dose
Population: All participants with ≥5 post-dosing samples available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years)
Number analyzed (Participants) | 9 | 5 | 4 | 8 | 6 | 6
L/hr | 2.30 (21.4) | 3.58 (26.2) | 4.68 (52.5) | 2.26 (29.4) | 3.43 (105) | 5.69 (24.1)

3. Primary Outcome: Apparent Volume of Distribution (Vz) of Sugammadex [Part A]
Description: The Vz of sugammadex, defined as the amount of drug administered relative to plasma concentrations, was determined in each Part A arm.
Time Frame: 2 minutes (min), 15 min, 30 min, 60 min, 4-6 hours (hrs), and 10 hrs post-dose
Population: All participants with ≥5 post-dosing samples available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years)
Number analyzed (Participants) | 9 | 5 | 4 | 8 | 6 | 6
Liters | 3.58 (21.3) | 6.65 (33.5) | 10.8 (34.8) | 4.00 (37.7) | 8.22 (82.9) | 12.3 (35.9)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Sugammadex [Part A]
Description: The Cmax of sugammadex, defined as the maximum plasma concentration, was determined in each Part A arm.
Time Frame: 2 minutes (min), 15 min, 30 min, 60 min, 4-6 hours (hrs), and 10 hrs post-dose
Population: All participants with ≥5 post-dosing samples available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years)
Number analyzed (Participants) | 9 | 5 | 4 | 8 | 6 | 6
µg/mL | 17.5 (33.1) | 32.2 (15.6) | 41.3 (85.8) | 47.1 (22.1) | 51.6 (69.2) | 61.9 (13.5)

5. Primary Outcome: Plasma Half-Life (t½) of Sugammadex [Part A]
Description: The t½ of sugammadex, defined as the time required for the plasma concentration to decrease to 50% of maximum, was determined in each Part A arm.
Time Frame: 2 minutes (min), 15 min, 30 min, 60 min, 4-6 hours (hrs), and 10 hrs post-dose
Population: All participants with ≥5 post-dosing samples available are included.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years)
Number analyzed (Participants) | 9 | 5 | 4 | 8 | 6 | 6
Hours | 1.15 [0.964 to 1.64] | 1.19 [1.01 to 1.71] | 1.49 [1.17 to 1.91] | 1.12 [0.922 to 1.78] | 1.56 [1.21 to 3.06] | 1.51 [1.20 to 1.91]

6. Primary Outcome: Percentage of Participants With ≥1 Adverse Event (AE) [Parts A and B]
Description: The percentage of participants with ≥1 AE(s) for up to 7 days after treatment was determined for each treatment group, pooled according to treatment received. An AE is defined as any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated.
Time Frame: Up to 7 days
Population: Each participant who received a dose of study drug is included.
Measure: Number; unit: Percentage of Participants
Groups:
- Parts A and B: Sugammadex 2 mg: All participants in Parts A and B who received sugammadex 2 mg are included in the analysis.
- Parts A and B: Sugammadex 4 mg: All participants in Parts A and B who received sugammadex 4 mg are included in the analysis.
Arm/Group | Part B: Neostigmine + (Glycopyrrolate or Atropine) | Parts A and B: Sugammadex 2 mg | Parts A and B: Sugammadex 4 mg
Number analyzed (Participants) | 34 | 51 | 191
Percentage of Participants | 97.1 | 78.4 | 74.9

7. Primary Outcome: Time to Recovery of Participant Train-of-Four (TOF) Ratio to ≥0.9 [Part B]
Description: The time to recovery of TOF ratio to ≥0.9 after administration of study intervention was determined for each Part B arm. The TOF ratio is the ratio of the magnitude of the fourth (T4) and first (T1) thumb twitches elicited by 4 electrical stimulations of the ulnar nerve, indicating the current degree of NMB as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Values closer to 1 indicate less NMB. Per protocol, the efficacy analysis is based on comparison of the Part B: Sugammadex 2 mg arm versus the Part B: Neostigmine + (Glycopyrrolate or Atropine) arm.
Time Frame: Up to 30 minutes post-dose
Population: All randomized participants in Part B who received ≥1 dose of study drug are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 33 | 169 | 34
Minutes | 1.6 (1.3) [1.3 to 2.0] | 1.9 (1.7) [1.7 to 2.2] | 7.5 (5.6) [5.6 to 10.0]
Statistical Analysis 1: Comparison: Part B: Sugammadex 2 mg/kg vs Part B: Neostigmine + (Glycopyrrolate or Atropine); Test type: Superiority; p < 0.0001, ANOVA; GM Ratio (SUG 2 mg / NEO + [GLY or ATR]) = 0.22, 95% CI 2-sided [0.16 to 0.32]

8. Secondary Outcome: Time to Recovery of Participant TOF Ratio to ≥0.7 [Part B]
Description: The time to recovery of TOF ratio to ≥0.7 after administration of study intervention was determined for each Part B arm. The TOF ratio is the ratio of the magnitude of the fourth (T4) and first (T1) thumb twitches elicited by 4 electrical stimulations of the ulnar nerve, indicating the current degree of NMB as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Values closer to 1 indicate less NMB.
Time Frame: Up to 30 minutes post-dose
Population: All randomized participants in Part B who received ≥1 dose of study drug are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 33 | 169 | 34
Minutes | 1.1 (0.9) [0.9 to 1.3] | 1.3 (1.1) [1.1 to 1.4] | 3.7 (2.9) [2.9 to 4.8]

9. Secondary Outcome: Time to Recovery of Participant TOF Ratio to ≥0.8 [Part B]
Description: The time to recovery of TOF ratio to ≥0.8 after administration of study intervention was determined for each Part B arm. The TOF ratio is the ratio of the magnitude of the fourth (T4) and first (T1) thumb twitches elicited by 4 electrical stimulations of the ulnar nerve, indicating the current degree of NMB as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Values closer to 1 indicate less NMB.
Time Frame: Up to 30 minutes post-dose
Population: All randomized participants in Part B who received ≥1 dose of study drug are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Part B: Sugammadex 2 mg/kg | Part B: Sugammadex 4 mg/kg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
Number analyzed (Participants) | 33 | 169 | 34
Minutes | 1.3 (1.1) [1.1 to 1.6] | 1.5 (1.3) [1.3 to 1.7] | 5.0 (3.8) [3.8 to 6.7]

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. All participants who received ≥1 dose of study drug are included.
Groups:
- Part B: Sugammadex 2 mg: For moderate NMB reversal, a single i.v. bolus of sugammadex (2 mg/kg) was given after final dose of neuromuscular blocking agent (NMBA; rocuronium or vecuronium) and within 2 minutes of the reappearance of a second twitch (T2) in response to TOF stimulations.
- Part B: Sugammadex 4 mg: For deep NMB reversal, a single i.v. bolus of sugammadex (4 mg/kg) was given after final dose of NMBA (rocuronium or vecuronium) and within 2 minutes of detection of a target of 1 to 2 post-tetanic counts and no response to TOF stimulations (TOF=0).
Arm/Group | Part A: Sugammadex 2 mg (2 to <6 Years) | Part A: Sugammadex 2 mg (6 to <12 Years) | Part A: Sugammadex 2 mg (12 to <17 Years) | Part A: Sugammadex 4 mg (2 to <6 Years) | Part A: Sugammadex 4 mg (6 to <12 Years) | Part A: Sugammadex 4 mg (12 to <17 Years) | Part B: Sugammadex 2 mg | Part B: Sugammadex 4 mg | Part B: Neostigmine + (Glycopyrrolate or Atropine)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5 | 0/4 | 0/10 | 0/6 | 0/6 | 0/33 | 0/169 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5 | 0/4 | 0/10 | 0/6 | 0/6 | 3/33 | 3/169 | 2/34
Other Adverse Events (participants affected / at risk) | 8/9 | 3/5 | 2/4 | 8/10 | 5/6 | 6/6 | 26/33 | 117/169 | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Sugammadex 2 mg (2 to <6 Years) (N=9) | Part A: Sugammadex 2 mg (6 to <12 Years) (N=5) | Part A: Sugammadex 2 mg (12 to <17 Years) (N=4) | Part A: Sugammadex 4 mg (2 to <6 Years) (N=10) | Part A: Sugammadex 4 mg (6 to <12 Years) (N=6) | Part A: Sugammadex 4 mg (12 to <17 Years) (N=6) | Part B: Sugammadex 2 mg (N=33) | Part B: Sugammadex 4 mg (N=169) | Part B: Neostigmine + (Glycopyrrolate or Atropine) (N=34)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Sugammadex 2 mg (2 to <6 Years) (N=9) | Part A: Sugammadex 2 mg (6 to <12 Years) (N=5) | Part A: Sugammadex 2 mg (12 to <17 Years) (N=4) | Part A: Sugammadex 4 mg (2 to <6 Years) (N=10) | Part A: Sugammadex 4 mg (6 to <12 Years) (N=6) | Part A: Sugammadex 4 mg (12 to <17 Years) (N=6) | Part B: Sugammadex 2 mg (N=33) | Part B: Sugammadex 4 mg (N=169) | Part B: Neostigmine + (Glycopyrrolate or Atropine) (N=34)
Bradycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 9 (9) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 10 (10) | 2 (2)
Palatal swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 20 (22) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 9 (9) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 1 (1) | 7 (7) | 3 (3) | 3 (3) | 22 (22) | 98 (109) | 24 (25)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03351608/Prot_SAP_000.pdf